CLINICAL TRIAL: NCT06082206
Title: Pectoral Nerve Block Versus Paravertebral Block In The Incidence of Chronic Pain After Mastectomy: A Randomized Clinical Trial
Brief Title: Pectoral Nerve Block Versus Paravertebral Block In The Incidence of Chronic Pain After Mastectomy:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pectoral N VS Paravertebral
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Paravertebral Block; Pectoral Nerve Block; Chronic Pain; Mastectomy; Lymphedema
MeSH Terms: conditions — Chronic Pain; Lymphedema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPVB Group (Experimental): Bupivacaine 0.25% 20 ml was injected between the costotransverse ligament and the parietal pleura.
  Interventions: Procedure: thoracic paravertebral block (TPVB)
- PECS Group (Experimental): bupivacaine 0.25% 10 ml
  Interventions: Procedure: PECS group

INTERVENTIONS:
Procedure: thoracic paravertebral block (TPVB) — Bupivacaine 0.25% 20 ml was injected between the costotransverse ligament and the parietal pleura.
  Arms: TPVB Group
Procedure: PECS group — entering the plane between the pectoralis minor muscle and serratus anterior muscle, and bupivacaine 0.25% 10 ml was deposited in this space
  Arms: PECS Group

SUMMARY:
Chronic pain after Mastectomy is frequent and an important healthcare priority because of its effect on quality of life. Although the association between the severity of acute pain after surgery and the likelihood of chronic pain is known, their causal relationship has not been clarified. Mastectomy, frequently done for the management of breast cancer, is associated with significant acute postoperative pain and limited shoulder movement.

DETAILED DESCRIPTION:
General anesthesia with postoperative NSAI D and opioids is a commonly used technique for postoperative analgesia after breast surgeries. Patients with mastectomy under general anesthesia commonly have pain in the axilla and upper limb that increases hospital stay, costs, and postoperative complications .Thoracic paravertebral block can be performed for analgesia after breast surgery. Ultrasound usage gave an accurate reading of the depth to the paravertebral space and can be used during the whole technique. Breast surgery is usually done with axillary dissection and can be done at single or multiple levels of thoracic paravertebral blocks .Thoracic paravertebral block is associated with multiple complications such as hypotension, pneumothorax, sympathetic block, central spread of local anesthesia or failed block which may cause limitations in the technique. The use of ultrasound in anesthesia increases the success rate of the block and decreases the incidence of variable complications .On the other hand, many interfascial plane blocks have been described. Pectoral nerve block (PECS) has been described as interfascial plane blocks and provide analgesic adjuvants for breast surgery with or without axillary dissection. The block was described as an injection of local anesthetic between the pectoralis major and minor muscles (PEC I) and between pectoralis minor and serratus anterior muscle (PEC 2) .

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I, II, or III female patients in the age group of 20-65 years
* with body mass index (BMI) of 25-35 who were undergoing mastectomy with or without axillary lymph node or sentinel lymph node dissection or partial mastectomy (sparing the skin, areola, and nipple) with axillary lymph node dissection

Exclusion Criteria:

* male sex; patient refusal,
* a life expectancy less than 2 yr;
* active malignant disease; pregnant or breastfeeding women;
* bilateral surgery; ipsilateral breast surgery in the past 3 yr;

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of chronic pain | 3 and 6 months
  The incidence of chronic pain, 0 to 10 Numerical Rating scale (NRS) 3 and 6 months after breast surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Simpson J, Ariyarathenam A, Dunn J, Ford P. Breast surgery using thoracic paravertebral blockade and sedation alone. Anesthesiol Res Pract. 2014;2014:127467. doi: 10.1155/2014/127467. Epub 2014 Aug 21. PMID 25214832